CLINICAL TRIAL: NCT02833779
Title: Trial to Compare the Effectiveness of Group Versus Individual Therapy on Alternate Days in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Marcos Sanchez Garcia, Registered physiotherapist, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSD
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Mobility

ARMS (2):
- Group Therapy Exercises (Active Comparator): Patients will be taught exercises in groups of six persons, on a daily basis for twelve sessions.
  Interventions: Other: Group exercises
- Individual Manual Therapy Exercises (Active Comparator): Patients will be taught the same exercises as in a Group 1, individually, and will receive manual therapy consisting of muscular and joint re-centering
  Interventions: Other: Individual exercises

INTERVENTIONS:
Other: Individual exercises
  Arms: Individual Manual Therapy Exercises
Other: Group exercises
  Arms: Group Therapy Exercises

SUMMARY:
Pathology of the rotator cuff and subacromial bursa is considered to be the principal cause of pain and symptoms arising from the shoulder. Physiotherapy specialists often disagree about which type of exercise is most appropriate. Manual Physiotherapy combined with guided exercise is a commonly applied clinical treatment, but no proof of its effectiveness has been shown. Clinical trials comparing results of treating subacromial syndrome of the shoulder with guided self-treatment and conventional physiotherapy yielded a slightly higher improvement, basically because patients suffered from chronic tendinitis and the treatment period lasted only two weeks. That is the reason why the investigators propose a long-term follow-up study and a more complete assessment of effectiveness of the exercise prescribed to improved this pathology.

Objectives:

* Assessment of effectiveness of two different types of treatment of subacromial syndrome of the shoulder.
* Comparison of effectiveness of both treatments in order to select that one yielding better results as the one to be applied as a routine practice.

Patients will be assigned one of the following treatments:

* Group 1: patients will be taught exercises in groups of six people, on a daily basis for twelve sessions.
* Group 2: patients will be taught the same exercise as Group 1, individually, and will receive manual therapy consisting of muscular and joint re-centering.

A modified version of the Constant scale will be used to assess mobility and pain shoulder.

ELIGIBILITY:
Inclusion Criteria:

* History of shoulder pain defined as at least 2 positive results in subacromial impingement tests.
* Self-perceived pain reported by the patient under clinical examination of the shoulder.
* A minimum of 90º mobility in flexion.

Exclusion Criteria:

* Luxation, a history of surgery, or evidence the current shoulder pain or other symptoms under cervical examination or other shoulder bone disease, except for acromioclavicular joint arthrosis.
* Patients were receiving other physiotherapy or rehabilitation treatments.
* Patients had been treated for SIS (subacromial impingement syndrome) with injection of anti-inflammatory or analgesic drugs in the last month.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The assessment of pain with a visual analogue scale. | Six Months
The mobility (joint range of motion) with a goniometer. | Six Months